CLINICAL TRIAL: NCT01799954
Title: A Phase 1 Double Blind Placebo-controlled Clinical Trial to Evaluate the Safety and to Compare the Priming Ability of NYVAC Alone Versus NYVAC + AIDSVAX® B/E, and DNA Alone Versus DNA + AIDSVAX® B/E When Followed by NYVAC + AIDSVAX® B/E Boosts in Healthy, HIV-1-uninfected Adult Participants
Brief Title: Evaluating the Safety and Priming Response of an HIV Vaccine Regimen in Healthy, HIV-Uninfected Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: HIV Vaccine Trials Network (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HVTN 096
Record Dates: First submitted 2013-02-22; First posted 2013-02-27 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2015-03

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Vaccines, DNA

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- NYVAC Prime / NYVAC + AIDSVAX® B/E Boost vs. Placebo (Other): This arm will evaluate the safety of and the body's immune response to a vaccine regimen consisting of a NYVAC vaccine prime and NYVAC + AIDSVAX® B/E boost. Twenty participants will get vaccines and 4 will get only placebos.
  Interventions: Biological: NYVAC-HIV-PT1; Biological: NYVAC-HIV-PT4; Biological: AIDSVAX® B/E; Biological: Placebo for DNA/NYVAC; Biological: Placebo for AIDSVAX(R) B/E
- NYVAC + AIDSVAX® B/E Prime / Boost vs. placebo (Other): This arm will evaluate the safety of and the body's immune response to a vaccine regimen consisting of priming and boosting with the vaccines NYVAC + AIDSVAX® B/E. Twenty participants will receive the vaccines and 4 will receive placebos. This arm will also be compared to arm 1 to see if the priming makes a difference in the body's immune response.
  Interventions: Biological: NYVAC-HIV-PT1; Biological: NYVAC-HIV-PT4; Biological: AIDSVAX® B/E; Biological: Placebo for DNA/NYVAC; Biological: Placebo for AIDSVAX(R) B/E
- DNA prime + NYVAC + AIDSVAX® B/E Boost vs. placebo (Other): This arm will evaluate the safety of and the body's immune response to a vaccine regimen consisting of a DNA vaccine priming and NYVAC + AIDSVAX® B/E boosting. Twenty participants will receive the vaccines and 4 will receive placebos. This arm will also be compared to arm 4 to see if the priming makes a difference in the body's immune response.
  Interventions: Biological: DNA-HIV-PT123; Biological: NYVAC-HIV-PT1; Biological: NYVAC-HIV-PT4; Biological: AIDSVAX® B/E; Biological: Placebo for DNA/NYVAC; Biological: Placebo for AIDSVAX(R) B/E
- DNA+AIDSVAX® B/E prime / NYVAC+AIDSVAX® B/E boost vs. placebo (Other): This arm will evaluate the safety of and the body's immune response to a vaccine regimen consisting of a DNA vaccine + AIDSVAX® B/E priming and NYVAC + AIDSVAX® B/E boosting. Twenty participants will receive the vaccines and 4 will receive placebos. This arm will also be compared to arm 3 to see if the priming makes a difference in the body's immune response.
  Interventions: Biological: DNA-HIV-PT123; Biological: NYVAC-HIV-PT1; Biological: NYVAC-HIV-PT4; Biological: AIDSVAX® B/E; Biological: Placebo for DNA/NYVAC; Biological: Placebo for AIDSVAX(R) B/E

INTERVENTIONS:
Biological: DNA-HIV-PT123 — 4 mg of DNA encoding clade C ZM96 Gag and gp140, CN54 Pol-Nef, administered intramuscularly (IM)
  Other Names: DNA Vaccine
  Arms: DNA prime + NYVAC + AIDSVAX® B/E Boost vs. placebo; DNA+AIDSVAX® B/E prime / NYVAC+AIDSVAX® B/E boost vs. placebo
Biological: NYVAC-HIV-PT1 — (along with NYVAC-HIV-PT4); ≥ 5x106 PFU encoding clade C ZM96 gp140 and ZM96 Gag and CN54 Pol-Nef, administered IM
Biological: NYVAC-HIV-PT4 — (along with NYVAC-HIV-PT1); ≥ 5x106 PFU encoding clade C ZM96 gp140 and ZM96 Gag and CN54 Pol-Nef, administered IM
Biological: AIDSVAX® B/E — 300mcg of subtype B (MN) HIV gp120 glycoprotein and 300mcg of subtype E (A244) HIV gp120 glycoprotein absorbed onto 600mcg of aluminum hydroxide gel adjuvant, administered IM.
Biological: Placebo for DNA/NYVAC — Sodium Chloride for injection, 0.9% administered IM
Biological: Placebo for AIDSVAX(R) B/E — 600 mcg of aluminum hydroxide adjuvant, administered IM

SUMMARY:
This study will evaluate the safety of and the body's immune response to experimental HIV vaccine regimens using different vaccine priming combination, and boosting with the vaccines NYVAC and AIDSVAX® B/E.

DETAILED DESCRIPTION:
Although multiple candidate HIV vaccines are being studied, there is not yet an effective preventive HIV vaccine. This study will test 4 experimental HIV vaccine regimens, each boosting with the NYVAC + AIDSVAX® B/E vaccine combination. Priming will be done with NYVAC or DNA vaccines, alone or in combination with AIDSVAX® B/E.

The study will enroll 96 healthy participants, ages 18 - 50 years. Participants will be randomly assigned to 1 of 4 groups. In each group, there will be 20 participants who receive the vaccine regimen and 4 receiving only placebo. Injections will take place at months 0, 1, 3, and 6.

All groups will enroll simultaneously. Enrollment will be restricted to a maximum of 2 participants per day, with no more than (1) participant in group 1 or 2 and (1) participant in group 3 or 4 until 20 participants have been enrolled with 5 in each group (4 vaccine recipients and 1 placebo recipient in each group). The HVTN 096 PSRT will review the safety and immune response data for the first 168 hours postvaccination on each of these participants, and will determine whether it is safe to proceed with full enrollment.

Total study duration will be 60 months: 18 months of clinic visits followed by annual health contacts to a total of 5 years after initial study injection. At the screening visit, participants will give a medical history and undergo a complete physical exam, cardiac symptom assessment (including ECG), urine collection, blood collection, interview, HIV test, and pregnancy test (for participants who were born female). On Days 0, 28, 84, and 168 participants will receive intramuscular (IM) vaccination (vaccine or placebo) into the right and left deltoids. On vaccination visits, participants will also undergo an abbreviated physical exam, cardiac symptom assessment, Social impact assessment, a pregnancy test (for participants who were born female), risk-reduction counseling, and blood collection. Immediately following vaccination, participants will remain in the clinic for observation for 30 minutes; participants will be given a post-vaccination symptom log and instructed on how to complete it. Follow-up visits will consist of a brief physical exam, blood collection, and interview; some follow-up visits may also consist of a urine collection, HIV test, or ECG. Optional mucosal secretion collection, if the participant agrees, will be done on days 0, 168, and 364.

The last clinic visit will be at Day 545; after this visit, participants will be contacted for annual health follow-up consisting of confirming vital status, collecting safety information, and reporting a new HIV diagnosis or a pregnancy. A clinic visit will only be required if HIV confirmatory testing is necessary.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 to 50 years
* Access to a participating HVTN CRS and willingness to be followed for the planned duration of the study
* Ability and willingness to provide informed consent
* Assessment of understanding: volunteer demonstrates understanding of this study; completes a questionnaire prior to first vaccination with verbal demonstration of understanding of all questionnaire items answered incorrectly
* Willing to be contacted annually after completion of scheduled clinic visits for a total of 5 years following initial study injection.
* Agrees not to enroll in another study of an investigational research agent
* Good general health as shown by medical history, physical exam, and screening laboratory tests
* Willingness to receive HIV test results
* Willingness to discuss HIV infection risks, amenable to HIV risk reduction counseling, and committed to maintaining behavior consistent with low risk of HIV exposure through the last required protocol clinic visit
* Assessed by the clinic staff as being at "low risk" for HIV infection
* Hemoglobin ≥ 11.0 g/dL for volunteers who were born female, ≥ 13.0 g/dL for volunteers who were born male
* White blood cell count = 3,300 to 12,000 cells/mm3
* Total lymphocyte count ≥ 800 cells/mm3
* Remaining differential either within institutional normal range or with site physician approval
* Platelets = 125,000 to 550,000/mm3
* Chemistry panel: ALT, AST, and alkaline phosphatase < 1.25 times the institutional upper limit of normal; creatinine <1.1x institutional upper limit of normal.
* Negative HIV-1 and -2 blood test: Non-US sites may use locally available assays that have been approved by HVTN Laboratory Operations.
* Negative Hepatitis B surface antigen (HBsAg)
* Negative anti-Hepatitis C virus antibodies (anti-HCV), or negative HCV polymerase chain reaction (PCR) if the anti-HCV is positive
* Normal urine:

  * Negative urine glucose, and
  * Negative or trace urine protein, and
  * Negative or trace urine hemoglobin (if trace hemoglobin is present on dipstick, a microscopic urinalysis with red blood cells levels within institutional normal range).
* Volunteers who were born female: negative serum or urine beta human chorionic gonadotropin (β-HCG) pregnancy test performed prior to vaccination on the day of initial vaccination
* Reproductive status: A volunteer who was born female must:

  * Agree to consistently use effective contraception (see Appendix B) for sexual activity that could lead to pregnancy from at least 21 days prior to enrollment through the last required protocol clinic visit. Effective contraception is defined as using any of the following methods:

    * Condoms (male or female) with or without a spermicide,
    * Diaphragm or cervical cap with spermicide,
    * Intrauterine device (IUD),
    * Hormonal contraception, or
    * Successful vasectomy in the male partner (considered successful if a volunteer reports that a male partner has [1] documentation of azoospermia by microscopy, or [2] a vasectomy more than 2 years ago with no resultant pregnancy despite unprotected sexual activity postvasectomy);
  * Or not be of reproductive potential, such as having reached menopause (no menses for 1 year) or having undergone hysterectomy, bilateral oophorectomy, or tubal ligation;
  * Or be sexually abstinent.
* Volunteers who were born female must also agree not to seek pregnancy through alternative methods, such as artificial insemination or in vitro fertilization until after the last required protocol clinic visit

Exclusion Criteria:

* Blood products received within 120 days before first vaccination
* Investigational research agents received within 30 days before first vaccination
* Intent to participate in another study of an investigational research agent during the planned duration of the HVTN 096/EV04 study
* Pregnant or breastfeeding
* HIV vaccine(s) received in a prior HIV vaccine trial. For volunteers who have received control/placebo in an HIV vaccine trial, the HVTN 096/EV04 PSRT will determine eligibility on a case-by-case basis.
* Non-HIV experimental vaccine(s) received within the last 5 years in a prior vaccine trial. Exceptions may be made for vaccines that have subsequently undergone licensure by the FDA. For volunteers who have received control/placebo in an experimental vaccine trial, the HVTN 096/EV04 PSRT will determine eligibility on a case-by-case basis. For volunteers who have received an experimental vaccine(s) greater than 5 years ago, eligibility for enrollment will be determined by the HVTN 096/EV04 PSRT on a case-by-case basis.
* Live attenuated vaccines other than influenza vaccine received within 30 days before first vaccination or scheduled within 14 days after injection (eg, measles, mumps, and rubella [MMR]; oral polio vaccine [OPV]; varicella; yellow fever)
* Influenza vaccine or any vaccines that are not live attenuated vaccines and were received within 14 days prior to first vaccination (eg, tetanus, pneumococcal, Hepatitis A or B)
* Allergy treatment with antigen injections within 30 days before first vaccination or that are scheduled within 14 days after first vaccination
* Immunosuppressive medications received within 168 days before first vaccination. (Not excluded: [1] corticosteroid nasal spray; [2] inhaled corticosteroids; [3] topical corticosteroids for mild, uncomplicated dermatitis; or [4] a single course of oral/parenteral corticosteroids at doses < 2 mg/kg/day and length of therapy < 11 days with completion at least 30 days prior to enrollment.
* Serious adverse reactions to vaccines including anaphylaxis and related symptoms such as hives, respiratory difficulty, angioedema, and/or abdominal pain. (Not excluded: a volunteer who had a nonanaphylactic adverse reaction to pertussis vaccine as a child.)
* Immunoglobulin received within 60 days before first vaccination
* Autoimmune disease
* Immunodeficiency
* Untreated or incompletely treated syphilis infection
* Clinically significant medical condition, physical examination findings, clinically significant abnormal laboratory results, or past medical history with clinically significant implications for current health. A clinically significant condition or process includes but is not limited to:

  * A process that would affect the immune response,
  * A process that would require medication that affects the immune response,
  * Any contraindication to repeated injections or blood draws,
  * A condition that requires active medical intervention or monitoring to avert grave danger to the volunteer's health or well-being during the study period,
  * A condition or process for which signs or symptoms could be confused with reactions to vaccine, or
  * Any condition specifically listed among the exclusion criteria below.
* Any medical, psychiatric, occupational, or other condition that, in the judgment of the investigator, would interfere with, or serve as a contraindication to, protocol adherence, assessment of safety or reactogenicity, or a volunteer's ability to give informed consent
* Psychiatric condition that precludes compliance with the protocol. Specifically excluded are persons with psychoses within the past 3 years, ongoing risk for suicide, or history of suicide attempt or gesture within the past 3 years.
* Current anti-tuberculosis (TB) prophylaxis or therapy
* Asthma exclusion criteria:

Asthma other than mild, well-controlled asthma. (Symptoms of asthma severity as defined in the most recent National Asthma Education and Prevention Program (NAEPP) Expert Panel report).

Exclude a volunteer who:

* Uses a short-acting rescue inhaler (typically a beta 2 agonist) daily, or
* Uses moderate/high dose inhaled corticosteroids, or
* In the past year has either of the following:

  * Greater than 1 exacerbation of symptoms treated with oral/parenteral corticosteroids;
  * Needed emergency care, urgent care, hospitalization, or intubation for asthma.

    * Diabetes mellitus type 1 or type 2, including cases controlled with diet alone. (Not excluded: history of isolated gestational diabetes.) Thyroidectomy, or thyroid disease requiring medication during the last 12 months
    * Hypertension:
* If a person has been found to have elevated blood pressure or hypertension during screening or previously, exclude for blood pressure that is not well controlled. Well-controlled blood pressure is defined as consistently ≤ 140 mm Hg systolic and ≤ 90 mm Hg diastolic, with or without medication, with only isolated, brief instances of higher readings, which must be ≤ 150 mm Hg systolic and ≤ 100 mm Hg diastolic. For these volunteers, blood pressure must be ≤ 140 mm Hg systolic and ≤ 90 mm Hg diastolic at enrollment.
* If a person has NOT been found to have elevated blood pressure or hypertension during screening or previously, exclude for systolic blood pressure ≥ 150 mm Hg at enrollment or diastolic blood pressure ≥ 100 mm Hg at enrollment.

  * BMI ≥ 40; ≤ 18; or BMI ≥ 35 with 2 or more of the following: age > 45, systolic blood pressure > 140 mm Hg, diastolic blood pressure > 90 mm Hg, current smoker, known hyperlipidemia
  * Bleeding disorder diagnosed by a doctor (eg, factor deficiency, coagulopathy, or platelet disorder requiring special precautions)
  * Malignancy (Not excluded: Volunteer who has had malignancy excised surgically and who, in the investigator's estimation, has a reasonable assurance of sustained cure, or who is unlikely to experience recurrence of malignancy during the period of the study)
  * Seizure disorder: History of seizure(s) within past three years. Also exclude if volunteer has used medications in order to prevent or treat seizure(s) at any time within the past 3 years.
  * Asplenia: any condition resulting in the absence of a functional spleen
  * History of hereditary angioedema, acquired angioedema, or idiopathic angioedema.

Hypersensitivity to eggs or egg products

* Subjects who have 2 or more of the following cardiac risk factors:

  * participant report of history of elevated blood cholesterol defined as fasting LDL > 160 mg/dL;
  * first degree relative (eg, mother, father, brother, or sister) who had coronary artery disease before the age of 50 years);
  * current smoker; or
  * body mass index (BMI) ≥ 35
* Electrocardiogram (ECG) with clinically significant findings, or features that would interfere with the assessment of myo/pericarditis, as determined by the contract ECG Lab, cardiologist, or study clinician including any of the following:

  * conduction disturbance (complete left or complete right bundle branch block or nonspecific intraventricular conduction disturbance with QRS ≥120 ms, any 2nd or 3rd AV block, or QTc prolongation [> 450 ms]);
  * significant repolarization (ST segment or T wave) abnormality;
  * significant atrial or ventricular arrhythmia;
  * frequent atrial or ventricular ectopy (eg, frequent premature atrial contractions, 2 premature ventricular contractions in a row);
  * ST elevation consistent with ischemia; or
  * evidence of past or evolving myocardial infarction
* History of myocarditis, pericarditis, cardiomyopathy, congestive heart failure with permanent sequelae, clinically significant arrhythmia (including arrhythmia requiring medication, treatment, or clinical follow-up

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2012-08; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of i) NYVAC prime with and without AIDSVAX® B/E plus NYVAC + AIDSVAX® B/E boosts; ii) DNA prime with and without AIDSVAX® B/E plus NYVAC + AIDSVAX® B/E boosts; | 7 days
  Local and systemic reactogenicity signs and symptoms, laboratory measures of safety, and adverse and serious adverse events. Signs and symptoms include pain, tenderness, and redness.
To evaluate and compare the body's immune response to 4 prime-boost regimens, comparing between: • NYVAC and NYVAC/AIDSVAX® B/E primes (Group 1 versus 2) • DNA and DNA/AIDSVAX® B/E primes (Group 3 versus 4) | 182 days
  HIV-specific binding antibody response as assessed by laboratory assay 2 weeks after the fourth vaccination
To evaluate and compare the durability of antibody response to different priming regimens when followed by two doses of NYVAC/AIDSVAX® B/E: • NYVAC and NYVAC/AIDSVAX® B/E primes (Group 1 versus 2) • DNA and DNA/AIDSVAX® B/E primes (Group 3 versus 4) | Days 182, 196, 273, 364, 455, 545
  HIV-specific antibody response as assessed at multiple timepoints between 2 weeks and 12 months after the last boost

SECONDARY OUTCOMES:
To evaluate and compare the body's immune response to priming regimens, comparing between: • NYVAC and NYVAC/AIDSVAX® B/E primes (Group 1 versus 2) • DNA and DNA/AIDSVAX® B/E primes (Group 3 versus 4) | Day 42
  HIV-specific antibody response as assessed 2 weeks after the second vaccination
To evaluate the body's immune response to different priming regimens when followed by two doses of NYVAC/AIDSVAX® B/E, comparing between: • Group 1 versus 2 • Group 3 versus 4 • Group 1 versus 3 • Group 2 versus 4 | Days 98 and 196
  * HIV-specific antibody responses 2 weeks after the third and fourth vaccinations
  * Antibody responses 2 weeks after the third and fourth vaccinations
  * Neutralizing antibodies magnitude and breadth against tier 1 and tier 2 HIV-1 2 weeks after the third and fourth vaccinations
  * Magnitude and frequency of HIV-specific T cell responses 2 weeks after the third and fourth vaccinations
To evaluate how long the immune response lasts in all 4 groups | Day 364
  HIV-1 specific antibodies and T-cell responses assessed through assays / bead array / flow cytometry 6 months post-last vaccination.
To evaluate the immune response to the 4 priming regimens | Day 42
  HIV-1 antibodies and T-cell responses assessed through assays, flow cytometry and/or multiplex bead array

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Pantaleo, MD, Study Chair — Centre Hospitalier Universitaire Vaudois Hospices (CHUV)
Locations (1):
- HVTN Clinical Research Site (HVTN CRS) ,, Lausanne, Switzerland

REFERENCES:
- [Derived] Moodie Z, Li SS, Giorgi EE, Williams LD, Dintwe O, Carpp LN, Chen S, Seaton KE, Sawant SS, Zhang L, Heptinstall J, Liu S, Grunenberg N, Tomaka F, Rerks-Ngarm S, Pitisuttithum P, Nitayaphan S, Ake JA, Vasan S, Pantaleo G, Frank I, Baden LR, Goepfert PA, Keefer M, Chirenje M, Hosseinipour MC, Mngadi K, Laher F, Garrett N, Bekker LG, De Rosa S, Andersen-Nissen E, Kublin JG, Lu S, Gilbert PB, Gray GE, Corey L, McElrath MJ, Tomaras GD. A polyvalent DNA prime with matched polyvalent protein/GLA-SE boost regimen elicited the most robust and broad IgG and IgG3 V1V2 binding antibody and CD4+ T cell responses among 13 HIV vaccine trials. Emerg Microbes Infect. 2025 Dec;14(1):2485317. doi: 10.1080/22221751.2025.2485317. Epub 2025 Apr 7. PMID 40190112
- [Derived] Pantaleo G, Janes H, Karuna S, Grant S, Ouedraogo GL, Allen M, Tomaras GD, Frahm N, Montefiori DC, Ferrari G, Ding S, Lee C, Robb ML, Esteban M, Wagner R, Bart PA, Rettby N, McElrath MJ, Gilbert PB, Kublin JG, Corey L; NIAID HIV Vaccine Trials Network. Safety and immunogenicity of a multivalent HIV vaccine comprising envelope protein with either DNA or NYVAC vectors (HVTN 096): a phase 1b, double-blind, placebo-controlled trial. Lancet HIV. 2019 Nov;6(11):e737-e749. doi: 10.1016/S2352-3018(19)30262-0. Epub 2019 Oct 7. PMID 31601541
- [Derived] Huang Y, Zhang L, Janes H, Frahm N, Isaacs A, Kim JH, Montefiori D, McElrath MJ, Tomaras GD, Gilbert PB. Predictors of durable immune responses six months after the last vaccination in preventive HIV vaccine trials. Vaccine. 2017 Feb 22;35(8):1184-1193. doi: 10.1016/j.vaccine.2016.09.053. Epub 2017 Jan 25. PMID 28131393